CLINICAL TRIAL: NCT02535052
Title: Investigating the Immune System in chrONIC Kidney Disease - the SONIC Study.
Brief Title: Investigating the Immune System in chrONIC Kidney Disease.
Acronym: SONIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Wellcome Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG_14-216
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Immune System Diseases; Chronic Kidney Disease
MeSH Terms: conditions — Immune System Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Peripheral Blood Mononuclear Cells, Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease (CKD) patients: Any gender, aged 65 years and over. Chronic kidney disease with eGFR between 15 and 60 ml/min. No immunological cause of kidney disease. Not immunosuppressed. To receive both seasonal influenza and pneumococcal polysaccharide vaccines as part of recommended clinical care.
  Interventions: Biological: Seasonal influenza and pneumococcal polysaccharide vaccines
- Healthy Control subjects: Any gender, aged 65 years and over. No known renal disease and eGFR 60ml/min or greater. Not immunosuppressed. To receive both seasonal influenza and pneumococcal polysaccharide vaccines as part of recommended clinical care.
  Interventions: Biological: Seasonal influenza and pneumococcal polysaccharide vaccines

INTERVENTIONS:
Biological: Seasonal influenza and pneumococcal polysaccharide vaccines — Vaccination

SUMMARY:
This study will investigate the function of the immune system in people with chronic kidney disease (CKD) compared to people with normal kidneys. The investigators will use standard vaccines - the seasonal flu vaccine and pneumococcal polysaccharide (Pneumovax) vaccine - to examine how the immune system responds to challenge. All subjects will receive these recommended vaccines as part of routine care. Blood and urine samples will be collected and tested at different time points to look at how the immune response develops to these vaccines and if there are any differences between people with CKD and those without. This will help us understand how CKD affects the function of the immune system.

DETAILED DESCRIPTION:
Compared to the general population, people with CKD are known to get more infections and are more likely to have complications from them. Protective measures such as vaccinations for common infections are not as effective in patients with CKD as they are in people with healthy kidneys. The reasons why this happens are not very clear. It is known that with increasing age, the body's immune defences are weakened, but it is not yet clear how different this is in older people with CKD compared to older people with healthy kidneys. Understanding how CKD affects the body's immune defence to new infections is vital in helping to prevent severe consequences from infection and make vaccination more effective for this group of people. This project aims to look at the function of immune cells in CKD patients and people with normal kidney function, together with their responses to clinically recommended vaccinations, including Pneumococcus (common pneumonia organism) and the influenza virus (the flu).

Study participants are invited to receive the clinically recommended seasonal influenza and pneumococcal polysaccharide vaccines during the seasonal influenza vaccination season (September - December), mirroring routine care they would receive in the community. Information on age, gender and pre-existing health problems, together with blood and urine samples will be collected from CKD patients for comparison with healthy volunteers at the following timepoints: day of vaccination, day 7 and 28 and 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* any gender
* aged 65 and over

Exclusion Criteria:

* Subjects who have had Pneumovax within last 5 years
* Subjects who have had current season's influenza vaccine
* CKD patients: eGFR less than 15ml/min or greater than 60ml/min, immune mediated cause of kidney disease.
* Healthy control subjects: known kidney disease, eGFR less than 60ml/min
* Subjects with comorbidities that are associated with an immunosuppressed state including, but not limited to, the following: Malignancy diagnosed within last 5 years except non-melanoma skin cancer; Solid organ (including kidney) or bone marrow transplant recipients; Blood borne viral infections: HIV, hepatitis B and C; Autoimmune disease e.g. vasculitis, rheumatoid arthritis; Previous splenectomy or asplenia from any other cause.
* Subjects currently taking any of the following immunosuppressive medications: Systemic corticosteroids e.g. prednisolone/dexamethasone; Chemotherapy agents e.g. cyclophosphamide, methotrexate, azathioprine; Biological therapies e.g. rituximab, infliximab, etanercept - including any administration within preceding 12 months.
* Subjects who have previously had a serious reaction to influenza vaccination, including anaphylaxis and Guillain-Barre Syndrome within 6 weeks of previous influenza vaccination
* Subjects who have a severe egg allergy (contraindication to influenza vaccination)
* Subjects who have previously had a serious reaction to the whole or any components of pneumococcal vaccination
* Subjects who have an active infection and/or are febrile on assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: CKD patients - individuals attending local tertiary care nephrology clinics.
  Healthy control subjects - individuals accompanying CKD patients to nephrology clinics or individuals invited to participate from Birmingham 1000 Elders Cohort.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving adequate humoral response to either vaccine | 28 days
  as assessed by vaccine-specific serum IgG levels

SECONDARY OUTCOMES:
Proportion of participants who maintain protective antibody titres to either vaccine at 6 months after vaccination | 6 months
  as assessed by vaccine-specific serum IgG levels
Relationship between eGFR and immune cell subsets following vaccination | 6 months
  investigatory outcome - will be assessed using flow cytometric techniques and established biochemical laboratory eGFR testing
Relationship between eGFR and reported infection rates | 6 months
  as assessed using established biochemical laboratory eGFR testing and participant reported infection-related events

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Harper, Principal Investigator — University of Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Wall N, Godlee A, Geh D, Jones C, Faustini S, Harvey R, Penn R, Chanouzas D, Nightingale P, O'Shea M, Richter A, Moss P, Cunningham A, Harper L. Latent Cytomegalovirus Infection and Previous Capsular Polysaccharide Vaccination Predict Poor Vaccine Responses in Older Adults, Independent of Chronic Kidney Disease. Clin Infect Dis. 2021 Aug 16;73(4):e880-e889. doi: 10.1093/cid/ciab078. PMID 33728434